CLINICAL TRIAL: NCT02763150
Title: Gestational Diabetes Prevention Program
Brief Title: Pre-pregnancy Lifestyle Intervention to Prevent the Recurrence of Gestational Diabetes in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CP-GDPP-trial
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Prevention
MeSH Terms: conditions — Diabetes, Gestational | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): Intervention group will receive a comprehensive, multicomponent weight loss intervention targeting diet, physical activity, and behavioral strategies.
  Interventions: Behavioral: Lifestyle intervention
- Health Promotion (Active Comparator): Health promotion group will receive education on healthy eating and activity before pregnancy.
  Interventions: Other: Health Promotion

INTERVENTIONS:
Behavioral: Lifestyle intervention — Intervention group will receive comprehensive behavioral weight loss program.
  Arms: Lifestyle Intervention
Other: Health Promotion — The health promotion group will receive education on healthy eating and activity
  Arms: Health Promotion

SUMMARY:
The overall purpose of this study is to determine the efficacy of a pre-pregnancy lifestyle intervention to reduce the recurrence of gestational diabetes mellitus in multiethnic women with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of gestational diabetes.
* BMI > 25 kg/m2
* Planning to have a baby in the next 1-3 years
* English or Spanish speaking

Exclusion Criteria:

* Age less than 18 years
* Women with Type 2 or Type 1 diabetes
* Current pregnancy
* Relocating in the next 2 years
* Medications that affect weight/diabetes
* Serious current physical disease
* History of eating disorders
* History of bariatric surgery
* Current problems with drug abuse
* Current treatment of a serious psychological disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Gestational Diabetes Mellitus | 26 weeks gestation

SECONDARY OUTCOMES:
Changes in maternal levels of fasting glucose | study entry, 16 weeks, 26 weeks gestation
Changes in maternal levels of fasting insulin | study entry, 16 weeks, 26 weeks gestation
Changes in maternal levels of systolic and diastolic blood pressure | study entry, 16 weeks, 26 weeks gestation
Changes in maternal levels of C-reactive protein | study entry, 16 weeks, 26 weeks gestation
Incidence of preeclampsia | Delivery
Incidence of cesarean delivery | Delivery
Weight changes | study entry, 16 weeks, 26 weeks gestation
Daily caloric intake | study entry, 16 weeks, 26 weeks gestation
Minutes per week of moderate physical activity | study entry, 16 weeks, 26 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (2):
- United States (2):
  - California Polytechnic State University, San Luis Obispo, California
  - Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available to outside investigators after the primary and secondary analyses are completed and in accordance with local institutional review board and NIH policies.

REFERENCES:
- [Derived] Phelan S, Jelalian E, Coustan D, Caughey AB, Castorino K, Hagobian T, Munoz-Christian K, Schaffner A, Shields L, Heaney C, McHugh A, Wing RR. Randomized controlled trial of prepregnancy lifestyle intervention to reduce recurrence of gestational diabetes mellitus. Am J Obstet Gynecol. 2023 Aug;229(2):158.e1-158.e14. doi: 10.1016/j.ajog.2023.01.037. Epub 2023 Feb 8. PMID 36758710
- [Derived] Phelan S, Jelalian E, Coustan D, Caughey AB, Castorino K, Hagobian T, Munoz-Christian K, Schaffner A, Shields L, Heaney C, McHugh A, Wing RR. Protocol for a randomized controlled trial of pre-pregnancy lifestyle intervention to reduce recurrence of gestational diabetes: Gestational Diabetes Prevention/Prevencion de la Diabetes Gestacional. Trials. 2021 Apr 7;22(1):256. doi: 10.1186/s13063-021-05204-w. PMID 33827659